CLINICAL TRIAL: NCT00458666
Title: Coagulation Parameters During Pregnancy in Amniotic Fluid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: CoagulationAmnioticFluid_CTIL
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-03

CONDITIONS: Pregnancy
Keywords: Amniotic fluid; D-dimer; coagulation; factor X activation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Amniotic fluid embolism is a rare devastating thromboembolic event, which is probably caused by the entrance of amniotic fluid (AF) to the maternal circulation. While AF contains coagulation activators, their role during pregnancy has not been elucidated. The current study aimed to evaluate coagulation parameters in AF during human pregnancy.

DETAILED DESCRIPTION:
Amniotic fluid embolism is a rare devastating thromboembolic event, which is probably caused by the entrance of amniotic fluid (AF) to the maternal circulation. While AF contains coagulation activators, their role during pregnancy has not been elucidated. The current study aimed to evaluate coagulation parameters in AF during human pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing amniocentesis during 15-35 weeks of gestation.

Exclusion Criteria:

* A history of venous thromboembolism
* Systemic disease i.e.; diabetes, hypertension, hypo or hyper-thyroidism,
* Anticoagulant treatment
* Abnormal embryo

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brenner, M.D, Principal Investigator — Rambam Health Care Campus; Arie Drugan, M.D, Study Chair — Rambam Health Care Campus
Locations (1):
- Dept of Obstetrics and Gynecology, Rambam-Health Care Campus, Haifa, Israel